CLINICAL TRIAL: NCT01808170
Title: Effect of Laparoscopic Ovarian Cystectomy of Endometrioma Versus Cyst Deroofing on Ovarian Reserve as Determined by Anti-mullerian Hormone and Antral Follicle Count: a Prospective Randomized Study.
Brief Title: Laparoscopic Ovarian Cystectomy of Endometrioma vs Deroofing and Ovarian Reserve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Mohamed S. Sweed lecturer of Obstetrics & Gynecology AinShams University., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05081985; m120984 (Other: AinShams University)
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Endometrioma
Keywords: Laparoscopy; AMH; AFC; Endometrioma; ovarian reserve; Ovarian cystectomy; ovarian cyst deroofing
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic ovarian cystectomy (Active Comparator): laparoscopic ovarian cystectomy will be performed on proliferative phase of menstrual cycle.Anti-mullerian hormone level measurement and estimation of antral follicle count will be done before surgery and will be repeated one month after surgery.
  Interventions: Procedure: Laparoscopic ovarian cystectomy
- laparoscopic cyst deroofing (Active Comparator): laparoscopic cyst deroofing will be performed on proliferative phase of menstrual cycle.Anti-mullerian hormone level measurement and estimation of antral follicle count will be done before surgery and will be repeated one month after surgery.
  Interventions: Procedure: laparoscopic cyst deroofing

INTERVENTIONS:
Procedure: Laparoscopic ovarian cystectomy — will be performed using video control under general anesthesia, pneumoperitoneum is induced by carbon dioxide, with three 5-mm trocars in the lower abdomen and a 10-mm intraumbilical main trocar, and we will use 5-mm scissors and graspers, and Ringer's lactate solution for irrigation. Before initiating ovarian surgery, the ovaries are completely freed with obtuse and sharp dissection.after a cleavage plane between the cyst wall and ovarian cortex is identified, the ovaries are pulled slowly and gently in opposite directions by means of two a traumatic grasping forceps. After removing the pseudo capsule from the abdominal cavity, selective minimal (15 watt) bipolar coagulation of bleeding is performed, without excessive coagulation of the surgical defect to avoid damaging the ovary.
  Arms: laparoscopic ovarian cystectomy
Procedure: laparoscopic cyst deroofing — will be performed using video control under general anesthesia, pneumoperitoneum is induced by CO2, with three 5-mm trocars in the lower abdomen and a 10-mm intraumbilical main trocar, and we will use 5-mm scissors and graspers, and Ringer's lactate solution for irrigation. Before initiating ovarian surgery, the ovaries are completely freed with obtuse and sharp dissection. after mobilizing the ovary, the contents of the cyst is removed with the suction-irrigator probe and the cavity is irrigated. The inside of the cyst is evaluated and the portion of ovarian cortex involved with endometriosis is removed. Small blood vessels from the ovarian bed and bleeding from the ovarian hilum can be controlled with bipolar electro coagulation (15 watt). Low-power bipolar coagulation applied to the inside wall of the redundant ovarian capsule
  Arms: laparoscopic cyst deroofing

SUMMARY:
The purpose of this study is to evaluate the impact of laparoscopic ovarian cystectomy versus laparoscopic cyst deroofing on ovarian reserve measured by serum levels of anti mullerian hormone and antral follicle count in patients with endometriomas.

DETAILED DESCRIPTION:
One of the major concerns about excision of endometriomas is their negative effect on ovarian reserve because of follicle loss, removal of endometriomas has been associated with poorer performance in IVF procedures, and decreased ovarian volumes have also been reported after surgery.Ovarian reserve is defined as the functional potential of the ovary which reflects the number and quality of the follicles left in the ovary, and is well-correlated with the response to ovarian stimulation using exogenous gonadotrophin. Over the years, various tests and markers of ovarian reserve have been reported; the static tests include serum markers, such as basal FSH, inhibin-B and anti-Mullerian hormone (AMH), and ultrasonographic markers, such as ovarian volume and antral follicle count.This study will include 122 patients aged between 18 and 35 years who have been diagnosed with endometrioma (unilateral or bilateral) and they are candidates for laparoscopic surgery. They will be selected according to inclusion and exclusion criteria.they will be randomized into two study groups, one study group will undergo laparoscopic ovarian cystectomy, the other study group will undergo laparoscopic cyst deroofing.AMH,AFC and ovarian volume will be measured pre-operative and post-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18-35 year
2. Regular menstrual cycles.
3. Endometrioma (unilateral or bilateral) diagnosed by transvaginal ultrasound with diameter ≥ 3 cm.

Exclusion criteria:

1. Any previous ovarian surgery.
2. Evidence of polycystic ovary syndrome according to Rotterdam criteria

   -Two of three of:
   * Oligo- or chronic anovulation.
   * Clinical and/or biochemical signs of hyperandrogenism.
   * Polycystic ovaries.
3. Evidence of premature ovarian failure diagnosed by follicle stimulating hormone level ≥40 IU/L
4. Any endocrinal disease affecting ovarian function e.g. thyroid dysfunction, hyperprolactinemia.
5. Previous hormonal medications e.g. oral contraceptive pills, gonadotropin-releasing hormone analogue within the last 3 months before surgery.
6. Any suspicious findings of ovarian malignant diseases diagnosed by transvaginal ultrasound.
7. Contraindication to surgery.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
comparison between the impacts of laparoscopic ovarian cystectomy and laparoscopic cyst deroofing on ovarian reserve as determined by alteration of AMH level in endometrioma patients. | 17 months

SECONDARY OUTCOMES:
comparison between the impacts of laparoscopic ovarian cystectomy and laparoscopic cyst deroofing on ovarian reserve as determined by antral follicle count estimation in endometrioma patients. | 17 months
comparison between the impacts of laparoscopic ovarian cystectomy and laparoscopic cyst deroofing on ovarian reserve as determined by ovarian volume estimation in endometrioma patients. | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K. Makled, M.D., Study Director — Assistant professor of Obstetrics & Gynecology, faculty of medicine, AinShams University; Mohamed S. Sweed, M.D., Principal Investigator — Lecturer Obstetics & Gynecolog, faculty of medicine, AinShams University; Neveen S. Mehanna, M.B.B.CH., Principal Investigator — AinShams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Sweed MS, Makled AK, El-Sayed MA, Shawky ME, Abd-Elhady HA, Mansour AM, Mohamed RM, Hemeda H, Nasr-Eldin EA, Attia NS, Eltaieb E, Allam H, Hussein A. Ovarian Reserve Following Laparoscopic Ovarian Cystectomy vs Cyst Deroofing for Endometriomas. J Minim Invasive Gynecol. 2019 Jul-Aug;26(5):877-882. doi: 10.1016/j.jmig.2018.06.022. Epub 2018 Sep 5. PMID 30193971